CLINICAL TRIAL: NCT02758249
Title: Anesthetic Effect on Immune Cell in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: KUH1160098
Record Dates: First submitted 2016-02-26; First posted 2016-05-02 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevoflurane (Active Comparator): patients under sevoflurane anesthesia
  Interventions: Drug: Sevoflurane
- propofol (Active Comparator): patients under propofol anesthesia
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Sevoflurane — patients are anesthetized by using sevoflurane inhalation
  Arms: sevoflurane
Drug: propofol — patients are anesthetized by using propofol infusion
  Arms: propofol

SUMMARY:
Anesthetics agents has an effect on immune response during the cancer surgery.This influence can regulatory to immune activity or cancer cell survival.

The purpose of this study is to prove the variation of immune cell activity between preoperative and postoperative period.

DETAILED DESCRIPTION:
The patients were allocated randomly to receive propofol or sevoflurane. Also, a total of 18ml of blood sample was obtained for total 3 times in consecutive order.

1. immediate before anesthesia induction
2. postoperative 1 hours
3. postoperative 24 hours

Immune cells isolation from patients peripheral blood mononuclear cells. Next, immune cell were co-culture with human cancer cell line (MCF-7) for 24 hours. investigation for immune cell or cancer cell survival by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* patient who was planned to undergo breast cancer surgery.

Exclusion Criteria:

* age < 20 years old
* history of hypersensitivity reaction in propofol or sevoflurane
* history of previous cancer
* patient with ongoing inflammation

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
immune cell (NK cell and CD8+ T cell) | up to 24 hours
  Patients blood sample are collect up to 24 hours postoperatively. These blood sample are collect in EDTA tube for NK cell and CD8+ T cell isolation from peripheral blood mononuclear cells (PBMCs). Isolation for NK cell, Ab stain with CD16 and CD56. Also, isolation for CD8+ T cell, Ab stain with CD8, that are purified from PBMCs, using FACSAria according to the manufacturer's protocol. These cell are culture with MCF-7 cancer cell line for 24 hours. After 24h, the degree of apoptosis of NK cell and CD8+ T cell was determined by flow cytometry. Suspension cell is NK cell or CD8+ T cell, these cells were harvest and washed with cell staining buffer. After washing, cell resuspended with Annexin-V binding buffer and stained with FITC-Annexin-V according to the manufacturer's protocol with analysis

SECONDARY OUTCOMES:
cancer cell (MCF-7) apoptosis | Baseline. postoperative 1 hours and 24 hours
  Patients blood sample are collect before and 1h after anesthesia induction and at 24h postoperatively. These blood sample are collect in EDTA tube for NK cell and CD8+ T cell isolation from peripheral blood mononuclear cells (PBMCs). Isolation for NK cell, Ab stain with CD16 and CD56. Also, isolation for CD8+ T cell, Ab stain with CD8, that are purified from PBMCs, using FACSAria according to the manufacturer's protocol. These cell are culture with MCF-7 cancer cell line for 24 hours. After 24h, the degree of apoptosis of cancer cell was determined by flow cytometry. Adherent cell is cancer cell, these cells were harvest and washed with cell staining buffer. After washing, cell resuspended with Annexin-V binding buffer and stained with FITC-Annexin-V according to the manufacturer's protocol with analysis

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D., Ph.D., Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim JA, Oh CS, Yoon TG, Lee JY, Lee SH, Yoo YB, Yang JH, Kim SH. The effect of propofol and sevoflurane on cancer cell, natural killer cell, and cytotoxic T lymphocyte function in patients undergoing breast cancer surgery: an in vitro analysis. BMC Cancer. 2018 Feb 7;18(1):159. doi: 10.1186/s12885-018-4064-8. PMID 29415668